CLINICAL TRIAL: NCT00780611
Title: Investigating the Improvement in 4D CT Images Using Audiovisual Biofeedback: An Intra-fraction and an Inter-fraction Evaluation.
Brief Title: Investigating the Improvement in 4D CT Images Using AV Biofeedback
Acronym: GCC0832
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Department of Radiation Oncology, Principal Investigator, University of Maryland, Baltimore
Other Study IDs: HP-00043968
Record Dates: First submitted 2008-10-24; First posted 2008-10-27 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Cancer of the Lung; Abdominal Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study will look at how tumors in the chest and abdomen move when you breathe. Your doctors are studying if extra 4D CT scans and instructions on how to breathe can help predict this type of movement and improve the accuracy of radiation treatment. 4D CT scans are approved by the FDA. A 4D CT scan is different from a regular CT because it moves slower and takes more pictures. It takes pictures of the way your body moves when you breathe. This gives doctors more pictures of your body so that they can match your pictures to the way you breathe.

In this study, instructions on how to breathe will be visual and audio. Visual instructions will be given to you on a computer screen. You will hear audio instructions through a speaker.

DETAILED DESCRIPTION:
JUSTIFICATION Among the various sites affected by cancer, statistics show that lung cancer is the leading cause of death among both men and women. One major reason for this is that the treatment of lung cancer has not improved drastically in the past few years. Lung tumors are also potentially difficult to treat with radiation therapy due the patients' respiration motion causing the tumor to be mobile.

A1) Detrimental effects of respiration motion Respiration motion affects all tumor sites in the thorax and abdomen, although the disease of most prevalence and relevance for radiotherapy is lung cancer. Many studies have been performed to study lung-tumor motion and methods to compensate for this motion during radiation treatment imaging, planning and delivery. The significance of the respiration motion compensation techniques is to reduce the mobility of the tumors and thereby reduce the dose to the surrounding normal structures. If no motion compensation methods are used then a margin must be added to ensure adequate coverage of the tumor. Large margins results in radiation delivered to a larger volume of critical structures.

A2) Compensation techniques Methods that reduce respiration induced intrafraction motion include active breathing control, voluntary breath-hold, deep inspiration breath-hold, respiratory gated techniques, and 4D or tumor-tracking techniques.1-6 Active breathing control and the deep inspiration breath hold involves the patient holding their breath. While these may improve the reproducibility of the position of the tumor within the lung, it is not feasible for all patients especially those that have a compromised respiratory function. Respiratory gating techniques involves turning on the beam during only a small window of the respiratory cycle. Thus respiratory gating reduces the intrafraction motion but does not totally eliminate it. During respiratory gating, since the beam is turned on and off based on the respiration signal, the treatment time may increase up to 35-40% compared to a regular treatment. Since the patient has to spend more time on the table, this could introduce more errors due to patient movement on the table. 4D or tumor tracking techniques has it own share of issues as is discussed in the following paragraph.

A3) During 4D radiotherapy (4DRT) delivery the tumor is continuously tracked with the radiation beam as they move throughout the respiratory cycle. The benefits of 4DRT are a reduction in dose to the healthy lung tissue and/or an increase in dose to the tumor. The gains from 4DRT are clinically measurable, though much development is needed in the various steps of 4DRT i.e. CT image acquisition, planning and delivery.

During 4D CT image acquisition, images are acquired during different respiration states of normal breathing.7-9 The quality of images acquired by using the 4D CT image acquisition is limited by patients respiration pattern. Since the images are sorted based on the patients respiration motion, any change in pattern could lead to the images being sorted to a different part of respiration. This effect is reflected as an artifact on the CT image.

Target volumes along with respiration motion can be determined by contouring the target in the various respiratory states thus obtaining a volume that encompasses an entire breathing cycle. The efficacy and accuracy of 4D CT will be maximized when patients breathe reproducibly. However it is well-known that respiration motion varies not only from one day to the next but also during one fraction.

A4) Effect of irregular breathing For 4D CT, minimizing the variation of patient breathing within a treatment fraction and from fraction to fraction, i.e., increasing the reproducibility of patient breathing, is important. Large variation in patient respiration motion and irregular breathing lead to artifacts in the CT images as shown in. However, respiration motion amplitude and period vary with time and from patient to patient because of various anatomic and physiologic factors.

A5) Possible solutions Biofeedback/coaching techniques are being increasingly embedded in the behavioral treatment of patients with lung disease such as chronic obstructive pulmonary disease, asthma, and cystic fibrosis. For respiratory gating, several studies suggest that verbal prompts improve respiration reproducibility. Kini et al.12 concluded that audio prompts improve the stability of respiration frequency of the patient but does not maintain the range of respiratory motion, whereas visual prompts control only the regularity of the displacement and the frequency is not reproducible. Based on the results of Kini et al.12, combined audio-visual biofeedback was devised to improve the reproducibility of respiration motion. Recently Neicu et al.13 described results of audio and visual prompting and demonstrated improvement in the efficacy of so-called synchronized moving aperture radiation therapy, using respiratory traces from single-patient and volunteer sessions.

George et al.14 concluded based on a 24-patient, multisession study that audio-visual biofeedback can significantly reduce residual motion variability for a given duty cycle, thus potentially improving the accuracy of respiratory-gating. From the results of this study it was seen that audio-visual biofeedback reduced motion by 0.5 cm (0.29 to 0.24 cm) for exhale breathing and 1.5 cm (0.46 to 0.36 cm) for inhale breathing.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old or older
* Patients undergoing a scan in the Department of Radiation Oncology for a thoracic or abdominal lesion(s) and identified as candidates for 4D CT.

Exclusion Criteria:

* Pregnant or breast-feeding women are excluded.
* Negative serum or urine pregnancy test prior to study entry is required. Once on the protocol, the patient will be advised and expected to implement an accepted and effective method of contraception such as oral contraceptives ('the pill'),intrauterine devices (IUD's), contraceptive implants under skin or contraceptive injections and condoms with foam.
* Patients who have difficulty lying flat on their back for extended periods of time will be excluded.

Ages: 18 Years to 86 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Abdominal & Thoracic malignancies who consent to recieving Radiation treatment at the University of Maryland, Baltimore, will be offered this protocol design.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2008-11; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of audio visual biofeedback for reducing artifacts for 4 -dimensional computer tomography (4DCT) | 8 scans over 3 days

SECONDARY OUTCOMES:
To evaluate improvement in acquisition of a 4D CT by using audio-visual biofeedback including acquisition procedure, tumor quality | 8 scans over 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Warren D'Souza, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Maryland, United States